CLINICAL TRIAL: NCT00776737
Title: Studies of Measures of Attention
Status: Completed | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090002; 09-DC-0002
Record Dates: First submitted 2008-10-18; First posted 2008-10-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-01-14

CONDITIONS: Attention Deficit Disorder; Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Disorder; Attention Deficit Hyperactivity Disorder; Computer Aided Learning; Attention Deficits; Healthy Volunteer; HV
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will compare two tests for attention deficit disorder (ADD) - the Test of Variables of Attention (TOVA) and the NIH Test of Attention - to see if they produce the same results. There are a number of problems with existing tests for ADD. For example, TOVA, the most commonly used test, operates only on older computers and has other problems as well. Because of these problems, NIDCD developed the new NIH Test of Attention. This study will determine if the new test is valid for ADD and how the performance on this test compares to the performance on the TOVA in the general population.

Healthy volunteers between 6 and 60 years of age who have no problems with sight or hearing and are not taking medication for ADD may be eligible for this study.

After a brief interview, participants take the first of the two study tests. On a second visit, they take the other of the two tests. Both tests ask the subject to respond to things they hear and see on a computer screen. Each test takes 30 to 45 minutes to complete. Some participants are asked to take the NIH Test of Attention a second time, on a third visit. Participants also take a 15- to 20-minute subtest of the Weschler Intelligence Test.

DETAILED DESCRIPTION:
Characterization of a new test of attention

Objective - The objective of this protocol is to provide normative data for population performance on the NIH Test of Attention, and to compare performance on this test with subjects' performance on the traditional Test of Variables of Attention (TOVA). The NIH Test of Attention has been developed to provide a modernized test that can be made available to researchers, clinicians, and educators free of charge.

Study population - A screened medically normal population sample containing adults and children of both sexes and all ethnicities without frank mental or sensory disabilities

Design - Subjects will be enrolled by outreach designed to gather a random population sample. Subjects will take the NIH Test of Attention at one testing session and the TOVA at another session. The population distribution of scores on the NIH Test of Attention will be ascertained, the standard descriptive statistics will be calculated, and the correlation of NIH Test of Attention scores with the TOVA scores in each subject will be measured. No individual identifying information will be gathered, and no test results will be provided back to subjects.

Outcome measures - The outcome will be measured by statistical tests for significant differences from the null hypothesis, which is that there is a difference in subject performance on the TOVA compared to the NIH Test of Attention. Mean, median, variance, and standard deviation of test scores will be calculated. Score distribution and Intra-class correlations will be quantified. Correlation of scores on the NIH Test of Attention with TOVA scores will be determined using Pearson's r.

ELIGIBILITY:
* INCLUSION CRITERIA:

Medically normal subjects, ages 6 to 60, who have a score of 25 or less on the Five Minute Hearing Test

EXCLUSION CRITERIA:

Subjects currently taking medication for ADD/ADHD, those with mental disability, hearing or vision impairment to the degree that subjects would fall under the criteria of the Americans with Disabilities Act. No vulnerable subjects will be enrolled, nor will subjects with an individual or family history of epilepsy.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2008-10-16; Study Completion 2011-01-14

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rowland AS, Lesesne CA, Abramowitz AJ. The epidemiology of attention-deficit/hyperactivity disorder (ADHD): a public health view. Ment Retard Dev Disabil Res Rev. 2002;8(3):162-70. doi: 10.1002/mrdd.10036. PMID 12216060
- [Background] Polanczyk G, Jensen P. Epidemiologic considerations in attention deficit hyperactivity disorder: a review and update. Child Adolesc Psychiatr Clin N Am. 2008 Apr;17(2):245-60, vii. doi: 10.1016/j.chc.2007.11.006. PMID 18295145
- [Background] Polanczyk G, Rohde LA. Epidemiology of attention-deficit/hyperactivity disorder across the lifespan. Curr Opin Psychiatry. 2007 Jul;20(4):386-92. doi: 10.1097/YCO.0b013e3281568d7a. PMID 17551354